CLINICAL TRIAL: NCT00447538
Title: Identifying Distress, Developmental and Behavioral Problems Among Toddlers, and Posttraumatic Distress Among Their Parents Following Continuous Exposure to Terrorism
Brief Title: Posttraumatic Symptoms Among Toddlers and Their Parents Following Exposure to Terrorism
Status: Completed | Type: Observational
Sponsor: Herzog Hospital (Other)
Collaborators: Picower Foundation (Other)
Other Study IDs: Rpat1CTIL
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The project utilize experience and knowledge gained from previous early childhood projects in NYC post 9/11 and Sderot. The overall goals are:

1. Identifying young children (under 6 years old) and their parents who are suffering from posttraumatic distress in the aftermath of the continuing conflict on Gaza border, Israel.
2. Increasing the capacity of local institutions to treat toddlers and families at risk.
3. Providing resilience -building services that strengthen the coping abilities of families and caregivers in response to continual terrorism.

DETAILED DESCRIPTION:
This project's aim is to identify psychological distress, build resilience among toddlers and their parents, and treat post traumatic stress disorder. The project components have consisted of a) using resilience-building interventions geared toward helping parents and daycare teachers deal with the stress engendered by the repeated emergency situations b) screening toddlers (24-48 months) for post traumatic distress utilizing new validated instruments c) referring highly symptomatic children and parents to dyadic treatment which focuses on observing the dynamics and interaction between parents and children before treatment intervention with the (more typically) mother/child.

Research into childhood trauma has clearly demonstrated that infants and children impacted by terrorism or with mothers who have suffered traumatic experiences are at very high risk for a multitude of long-term emotional disorders. Mothers suffering the effects of Post Traumatic Stress Disorders (PTSD) have difficulty providing the emotional holding environment and relational foundation necessary for healthy attachment and bonding. An anxious or traumatized mother will have difficulty soothing her child if she herself is in a state of emotional and physical hyper-arousal.

The project is aimed at identifying children who are suffering from posttraumatic distress and increasing capacity to provide treatment for them and for their caretakers. The project will be implemented in Sderot. Professional staff (teachers, nurses and aides) will be trained to conduct a systematic short screening in order to identify families with babies, toddlers and young children suffering from, or at risk for post-traumatic stress disorder.

The elements of the project will consist of:

A. Screening of young children and implementation of treatment The screening will consist of a short interviews with parents conducted by trained professional about exposure to traumatic events and resulting post-traumatic specific symptoms among the toddlers and their parents.

B. Workshops for parents, teachers, nurses The knowledge and skills of preschool teachers and nurses working in all our projects sights as well as parents will be increased by providing training regarding the impact of war related trauma on preschool children. Workshops will better equip teachers, nurses and parents with knowledge about the emotional impact of trauma on young children and will increase the skills to help preschool children contain emotional distress as well as to help them in coping with the emotional consequences of trauma exposure.

C. Treatment Interventions Dyadic treatment involving parents and children is aimed at increasing the attunement of parents to their toddlers and their needs in times of crises. Local practitioners in Sderot will received specialized training in this methodology by a child trauma specialist from Mount Sinai Medical Center in New York. The effectiveness of the dyadic treatment will be evaluated.

D. Evaluation of treatment Evaluation of treatment efficacy (dyadic treatment) will be assessed by pre and post interviews that will be conducted by trained professionals with all parents participating in the dyadic treatments in each of the three cities.

ELIGIBILITY:
Inclusion Criteria:

* Families with children between 24-48
* Families living in Sderot, Israel

Exclusion Criteria:

* Children with severe developmental problems

Ages: 24 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300
Dates: Start 2005-11; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Pat-Horenczyk, Ph.D, Principal Investigator — Israel Center for the Treatment of Psychotrauma
Locations (1):
- Sderot, Sderot, Israel